CLINICAL TRIAL: NCT05253248
Title: Development of an Optimal Micronutrient Reference Range for Adults
Acronym: OMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Konstantinos Gerasimidis (Other)
Responsible Party: Sponsor-Investigator, Dr Konstantinos Gerasimidis, Professor, University of Glasgow
Organization: University of Glasgow (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 200180119
Record Dates: First submitted 2022-01-13; First posted 2022-02-23 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Micronutrients Reference Interval; Micronutrients Normal Range

STUDY DESIGN:
Intervention Model Description: This is an open-label micronutrient supplementation trial in healthy adult volunteers. We are planning to supplement healthy adult volunteers, once a day, with a standard over-the-counter multivitamin supplement for a period of 30 consecutive days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy adults (Experimental): We are planning to supplement healthy adult volunteers, once a day, with a standard over-the-counter multivitamin supplement for a period of 30 consecutive days. Supplementation will provide the daily dietary recommendations of micronutrients, as these are established by the Department of Health, on top of the participant's free diet. Supplementation aims to correct any subclinical deficiencies the participants might have particularly those which are common in the general community. In the UK, a typical example is Vitamin D, due to lack of sunshine and selenium (a geochemical) whose content in the UK soil is depleted and therefore intake is often below the recommendations.
  Fasted blood and urine samples will be collected before, and again two-to-three days, post-supplementation.
  Interventions: Dietary Supplement: OMIS

INTERVENTIONS:
Dietary Supplement: OMIS — This is an open-label micronutrient supplementation trial in healthy adult volunteers. We are planning to supplement healthy adult volunteers, once a day, with a standard over-the-counter multivitamin supplement for a period of 30 consecutive days.

SUMMARY:
This study aims to develop optimal micronutrient reference intervals from blood samples collected from "ideal" healthy adults and following micronutrient supplementation to minimise the chance of subclinical deficiencies.

DETAILED DESCRIPTION:
Vitamins, minerals and trace elements, collectively referred to us as micronutrients, are important enzyme co-factors and co-enzymes, antioxidants and gene transcription factors. Most micronutrients are provided to the body through the diet however the body can produce some of them, including vitamin D, vitamin K and niacin. Micronutrients are needed in much smaller amounts than the macronutrients.

Vitamins have diverse biochemical functions, including cellular growth and differentiation, and organ and immune function. Minerals are inorganic substances which are involved in nerve and muscle function, enzymatic systems and bone. Adequate dietary vitamin and mineral intake is crucial, as deficiencies have been associated with a number of specific and non-specific symptoms which lead to loss of body homeostasis and disease onset. Beyond a suboptimal dietary intake, in illness, the aetiology of micronutrient deficiencies can be multifactorial and include malabsorption, excessive losses, increased nutrient requirements and drug-nutrient interactions.

There is continuous interest in the role of the micronutrients; both from a public health point of view, to prevent disease onset, and from a clinical practice perspective to monitor and treat deficiencies and optimise clinical outcomes. This interest stems from our increasing understanding in the biological roles of these nutrients, findings from epidemiological research, and the public interest on the potential health promoting benefits of these nutrients, as these are often portrayed to them by the commercial manufacturers of such supplements. It is also a common outcome that hypotheses generated from association studies and nutritional epidemiology are not replicated by intervention studies particularly when the latter ones aim to correct reduced blood concentrations of micronutrients or suboptimal intakes. These counterintuitive findings can be explained by other, often unknown, confounding factors that explain the relationship between the micronutrient status in the body and health or clinical outcomes, but also due to the fact that in several of these previous studies the methodology applied to assess the body micronutrient status in patient or population groups was insufficient or interpretation of the assessment outcomes were not reflective of the true micronutrient status of the body. From a clinical practice perspective there are five fundamental reasons why assessment of micronutrients is important: a) confirm the clinical manifestation of micronutrient deficiencies or toxicity; b) to screen and identify those at risk of micronutrient deficiencies or toxicity and refer them for further assessment; c) to prevent under or over-supplementation and its effects on patients prognosis; d) to supplement and potentially to improve the clinical outcomes of a patients with acute or chronic illness; e) to reduce health care associated expenditure from un-necessary use of resources to assess micronutrient status and from un-necessary interventions to correct non-existing deficiencies.

The mainstream approach to assess the micronutrient status of an individual, in-vivo, is the direct measurement of a micronutrient or its derivative concentration in biological fluids, mostly blood. However, there are several limitations with the use of laboratory biomarkers in ascertaining the micronutrient status of an individual. Development of blood micronutrient references for adults and children rely often on 95% confidence intervals established from measurements in samples drawn from the general population. Contrary to the concept of the new WHO centile growth charts, which describe the optimal pattern of growth for children, rather than the prevailing pattern in a population which is likely to be affected by environmental factors, there are no such standards for assessment of micronutrient status. Several of the micronutrient reference intervals used in health services and laboratories, particularly for the less commonly measured micronutrients (e.g. trace elements and B complex vitamins), are derived from very small convenience samples of essentially healthy individuals. It is therefore possible that these values are based on selective populations, and do not represent the distribution of the biomarker in the population and most importantly it may be based on populations in areas where there is a subclinical micronutrient insufficiency epidemic in the general population, (e.g. Vit D or Selenium in Scotland). As a result, use of such reference ranges may mask deficiency in an individual and underestimate the proportion of subjects with micronutrient deficiencies in a diseased population.

In human, a highly complex system also regulates redistribution of micronutrients in the presence of illness. It is believed that this system ensures that there is the right concentration of each micronutrient in the right tissue or body fluid at the various phases of the illness. The mechanisms behind these effects include uptake of nutrients to other tissues, shifts in vascular fluids and capillary permeability, loss of nutrient carrier protein, including serum albumin and lipoproteins and increased urinary excretion. As a result of these effects the blood concentration of several micronutrients will be affected, regardless of the actual body stores. A substantial amount of research shows that acute and chronic illness will affect blood micronutrient concentrations assayed in plasma with those measured in erythrocytes affected less or remain unaffected . Plasma concentrations of several nutrition-related biomarkers are known to be affected by inflammatory response, including vitamins retinol, C, B6, C, E and D, carotenoids, ferritin, zinc, copper and selenium. Where the nutrient or metabolite is a nutritional biomarker a depression in its concentrations will result in an overestimate of a deficiency. In contrast, where the biomarker is increased, as the results of an inflammatory illness, such as in infection and trauma, and as in the case of plasma ferritin and caeruloplasmin concentrations, this will result in an underestimate of iron and copper deficiency.

In conclusion, there are two unmet needs this proposal will try to address:

1. First, to develop optimal micronutrient reference ranges to overcome the inherent limitations of the existing ones.
2. Second, to develop novel, surrogate biomarkers, such as measurements in erythrocytes and other functional markers, whose levels remain uninfluenced by inflammatory diseases.

This study aims to develop optimal micronutrient reference intervals from blood samples collected from "ideal" healthy adults and following micronutrient supplementation to minimise the chance of subclinical deficiencies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (18 to 65 y) with BMI (18.5 to 27)
* Stable weight (±2kg)
* Non-smokers
* No regular medication
* Alcohol consumption less than 14 units per week
* on an unrestricted diet, and who live in postcodes belonging to the upper two quintiles of the Scottish Index of Multiple Deprivation (SIMD) and who are likely to have a diet close to the national recommendations established by Department of Health.

Exclusion Criteria:

* Individuals on restricted diets
* On intentional or unintentional weight loss
* overweight and obese (BMI > 27 kg/m2)
* Vegetarians
* Vegans
* Smokers
* Regular alcohol drinkers (>14 units per week)
* Those with special dietary requirements, food intolerances and on regular medication or nutrient supplements.
* Patients with mild conditions (i.e. conditions not requiring regular hospital, GP visits)
* Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Micronutrient reference centiles and reference intervals | Baseline
  Manganese, plasma zinc, plasma copper, plasma selenium, vit A, vit K, vit E, vit C, vit B1, vit B2, vit B6 and RBC selenium concentration will measured in Scottish Trace Element and Micronutrient Diagnostic and Research Laboratory using their routine methods. New micronutrient reference centiles for manganese, plasma zinc, plasma copper, plasma selenium, vit A, vit K, vit E, vit C, vit B1, vit B2, vit B6 and RBC selenium will be plotted on R using the GAMLSS package. 95% confidence intervals for mentioned above nutrients, representing the status of 95% of our population, will be calculated.
Differences | 33 days
  comparison between micronutrient status of the participants at baseline and the effect of supplementation will be calculated using paired t-tests.

SECONDARY OUTCOMES:
Micronutrients concentration and age | Baseline
  Correlation between micronutrients concentration and age
Micronutrients intake and concentration | Baseline
  Correlation between micronutrients intake and micronutrients concentration
Comparison of micronutrients concentration between Female and Male | 33 days
  Comparison of micronutrients concentration between Female and Male before and after Supplementation
Micronutrients concentration and body mass index | 33 days
  Correlation between micronutrients concentration and body mass index
Micronutrients concentration and lean mass index | 33 days
  Correlation between micronutrients concentration and lean mass index

CONTACTS AND LOCATIONS:
Locations (1):
- Maha Alik Al Fify, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No